CLINICAL TRIAL: NCT04387786
Title: Nebulized In-line Endotracheal Dornase Alfa and Albuterol Administered to Mechanically Ventilated COVID-19 Patients: A Case Series
Brief Title: Dornase Alfa Administered to Patients With COVID-19 (DACOVID)
Acronym: DACOVID
Status: Completed | Type: Observational
Sponsor: Feinstein Institute for Medical Research (Other)
Collaborators: Cold Spring Harbor Laboratory (Other)
Responsible Party: Principal Investigator, Betsy J Barnes, Investigator/Professor, Feinstein Institute for Medical Research
Organization: Northwell Health (Other)
Other Study IDs: 216
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; Mechanical Ventilation
MeSH Terms: conditions — COVID-19 | interventions — dornase alfa; Albuterol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Dornase Alfa — nebulized in-line endotracheal dornase alfa co-administered with albuterol
  Other Names: albuterol

SUMMARY:
Mechanically ventilated patients with coronavirus disease 2019 (COVID-19) have a mortality of 24-53%, in part due to distal mucopurulent secretions interfering with ventilation. Dornase alfa is recombinant human DNase 1 and digests DNA in mucoid sputum. Nebulized dornase alfa is FDA-approved for cystic fibrosis treatment. DNA from neutrophil extracellular traps (NETs) contributes to the viscosity of mucopurulent secretions. NETs are found in the serum of patients with severe COVID-19, and targeting NETs reduces mortality in animal models of acute respiratory distress syndrome (ARDS). Thus, dornase alfa may be beneficial to patients with severe COVID-19-acting as a mucolytic and targeting NETs.

DETAILED DESCRIPTION:
Demographic, clinical data, and outcomes were collected from the electronic medical records of five mechanically ventilated patients with COVID-19-including three requiring veno-venous extracorporeal membrane oxygenation (VV-ECMO)-treated with nebulized in-line endotracheal dornase alfa co-administered with albuterol (used to increase delivery to the alveoli), between March 31 and April 24, 2020. Data on tolerability and responses, including longitudinal values capturing respiratory function and inflammatory status, were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients with COVID-19

Exclusion Criteria:

* healthy, non-ventilated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Number of participants discharged from the intensive care unit (ICU) | 2 months
  discharge from ICU will be determined from the enterprise health record reporting database
Number of participants who survived COVID-19 | 2-4 months
  survival will be determined from the enterprise health record reporting database

SECONDARY OUTCOMES:
Mean change in FiO2 | 2 months
  fraction of inspired oxygen requirements will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Betsy J Barnes, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Insitute for Medical Research at Northwell Health, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
study will be published and data will be made available
Supporting Information: CSR
Time Frame: 3-6 months
Access Criteria: de-identified data

REFERENCES:
- [Background] Barnes BJ, Adrover JM, Baxter-Stoltzfus A, Borczuk A, Cools-Lartigue J, Crawford JM, Dassler-Plenker J, Guerci P, Huynh C, Knight JS, Loda M, Looney MR, McAllister F, Rayes R, Renaud S, Rousseau S, Salvatore S, Schwartz RE, Spicer JD, Yost CC, Weber A, Zuo Y, Egeblad M. Targeting potential drivers of COVID-19: Neutrophil extracellular traps. J Exp Med. 2020 Jun 1;217(6):e20200652. doi: 10.1084/jem.20200652. PMID 32302401